CLINICAL TRIAL: NCT00490321
Title: Evaluation of the VentrAssistTM Left Ventricular Assist Device for the Treatment of Advanced Heart Failure - Destination Therapy
Brief Title: VentrAssistTM LVAD for the Treatment of Advanced Heart Failure - Destination Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ventracor (Industry)
Collaborators: International Center for Health Outcomes and Innovation Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLP 12082
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: End-stage Heart Failure; Cardiomyopathies
Keywords: VentrAssistTM; LVAD; End-stage heart failure; Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: VentrAssistTM Left Ventricular Assist Device

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of LVADs in providing long-term circulatory support for patients who have chronic stage D heart failure and are ineligible for a heart transplant.

This is a multi-center, prospective, randomized, controlled clinical trial, which is comprised of two independent modules.

DETAILED DESCRIPTION:
Currently, patients with Stage D heart failure who are not transplant candidates are treated with a spectrum of therapies, including specialized medical management as well as mechanical support with an LVAD approved by FDA for destination therapy. However, there is substantial variation in the therapeutic approaches employed to treat these patients, with relatively low numbers of patients receiving DT LVAD therapy to date. Therefore, the VentrAssist DT trial is designed to provide maximal flexibility to the investigators/clinicians to incorporate their clinical judgment in managing these complex patients.

ELIGIBILITY:
Inclusion Criteria (The following are general criteria; detailed criteria are included in the study protocol):

* Eligible for either the VentrAssist or an FDA-approved DT LVAD
* LVEF <=25%
* Stage D heart failure
* Ineligible for cardiac transplantation
* Treated with standard heart failure therapy

Exclusion Criteria (The following are general criteria; detailed criteria are included in the study protocol):

* Contraindication to LVAD implantation
* Contraindication to anticoagulant or anti-platelet agents.
* Pre-existing mechanical circulatory support other than intra-aortic balloon pump
* Therapy with an investigational intervention at the time of screening
* A condition, other than heart failure, which would limit survival to less than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2007-06; Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Module A: Survival without a disabling stroke.
Module B: A composite endpoint of disabling stroke-free survival without device replacement or repair due to failure of the device to provide adequate circulatory support.

SECONDARY OUTCOMES:
•Safety •Functional Status and Hospitalizations •Quality of Life and Neurocognitive Assessment

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - University of Alabama, Birmingham, Alabama
  - Mayo Clinic, Phoenix, Arizona
  - University of Florida, Gainesville, Florida
  - Jackson Memorial, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - St. Vincent's, Indianapolis, Indiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Mount Sinai Hospital, New York, New York
  - Columbia University, New York, New York
  - Rochester Medical Center University, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Methodist Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Fairfax (Inova) Hospital, Falls Church, Virginia
  - University of Washington, Seattle, Washington
  - Sacred Heart Medical Center, Spokane, Washington
  - University of Wisconsin Hospital, Madison, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin